CLINICAL TRIAL: NCT02075281
Title: A 20-week, Double Blind, Randomized, Placebo Controlled, Parallel Group Trial to Assess the Safety and Efficacy of HM11260C on Body Weight in Obese Subjects Without Diabetes
Brief Title: Effect of LAPS-Exendin on Body Weight in Obese Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-EXC-205
Record Dates: First submitted 2014-02-25; First posted 2014-03-03 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- HM11260C (Experimental): HM11260C 4 mg weekly sc injection
  Interventions: Biological: HM11260C
- Placebo (Placebo Comparator): Placebo weekly sc injection
  Interventions: Biological: Placebo
- HM11260C 6 mg/week (Experimental): HM11260C 6 mg weekly sc injection
  Interventions: Biological: HM11260C
- HM11260C 6 mg/biweekly (Experimental): HM11260C 6 mg biweekly sc injection
  Interventions: Biological: HM11260C
- HM11260C 8 mg/biweekly (Experimental): HM11260C 8 mg biweekly sc injection
  Interventions: Biological: HM11260C

INTERVENTIONS:
Biological: HM11260C — Glucagon-like peptide-1 analogue
  Arms: HM11260C; HM11260C 6 mg/biweekly; HM11260C 6 mg/week; HM11260C 8 mg/biweekly
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the optimal dose and regimen of HM11260C, in combination with a hypocaloric diet, to reduce weight in obese subjects who are otherwise considered in stable health.

DETAILED DESCRIPTION:
Phase 2 study

ELIGIBILITY:
1. Inclusion Criteria:

   * Age: 18 years to 65 years
   * Genders: male and female
   * healthy obese population
   * non-diabetes
   * stable body weight for at least 3 months prior to screening
2. Exclusion Criteria

   * Pregnant or nursing (lactating) women
   * Drug-induced obesity
   * Diabetes mellitus (type 1, 2, and other)
   * Previous surgical treatment for obesity
   * Any known history of severe gastrointestinal (GI) disease or intolerance
   * Known history of pancreatitis with presence of raised serum amylase and lipase
   * History of suicide attempts or recent history (within 2 years prior to screening) of major depression, anxiety, or other psychiatric disease requiring treatment with prescription medication including selective serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitor s (SNRIs), antipsychotics, and lithium.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 297 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in body weight at 20 weeks | 20 weeks from baseline

SECONDARY OUTCOMES:
Number of participants with adverse event | during 20 weeks of treatment and follow-up period
Change from baseline in HbA1c and fasting plasma glucose level at 20 week | 20 weeks from baseline
Change from baseline in blood lipid profile (e.g., cholesterol, and LDL-C level) at 20 week | 20 weeks from baseline
  Cholesterol level, LDL-C level

OTHER OUTCOMES:
Change from baseline in waist circumference at 20 week | 20 weeks after baseline
Change from baseline in β-cell function at 20 week | 20 week from baseline
  homeostatic model assessment

CONTACTS AND LOCATIONS:
Overall Officials: Hanmi pharmaceuticals Hanmi pharmaceuticals, Principal Investigator — Hanmi pharmaceuticals
Locations (1):
- Hanmi pharmaceutical, Los Angeles, California, United States